CLINICAL TRIAL: NCT01246024
Title: Influence of Hypoxia on Electroretingraphy (ERG) Measurements
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Prof. Dr. med. Florian Gekeler, Centre for Ophthalmology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: THS0001
Record Dates: First submitted 2010-11-22; First posted 2010-11-23 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: ERG Under Hypoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypoxia (Experimental)
  Interventions: Device: ERG

INTERVENTIONS:
Device: ERG — scotopic and photopic ERG

SUMMARY:
To investigate the influence of induced hypoxia on the ERG.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* under 18 and over 80 years, respiratory diseases, cataracta and corneal hazes, myopia more than 6 dpt, hyperopia more than 3 dpt, allergy for any topical anesthetics in ophthalmology, photic epilepsy, asthma bronchiale.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Electroretingraphy Measurements | 01.02.2011-01.06.2011

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Ophthalmology, Tübingen, Germany